CLINICAL TRIAL: NCT03498560
Title: Examining the Association Between Pre-existing Sleep Disturbance and Postoperative Delirium
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Oluwaseun Johnson-Akeju, MD, MMSc, Associate Professor of Anaesthesia, Massachusetts General Hospital
Other Study IDs: 2018P000480
Record Dates: First submitted 2018-04-05; First posted 2018-04-13 (Actual); Results first posted 2020-09-04 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MGH Surgery Patients: PSG data will be collected, and delirium assessments conducted, on patients undergoing surgery at MGH.
  Interventions: Device: PSG

INTERVENTIONS:
Device: PSG — PSG data to be collected on the night before surgery to establish level of preexisting sleep disturbance.

SUMMARY:
The investigators are performing this research study to understand the role of sleep disturbance on the incidence/severity of delirium after surgery. The investigators will study the brain using a polysomnography device (PSG), which records the brain's electrical activity during sleep.

DETAILED DESCRIPTION:
During this study, PSG recordings will be collected and a sleep questionnaire will be administered to participants on the night before surgery in order to establish level of preexisting sleep disturbance. Delirium assessments will be conducted during the postoperative period. On postoperative days 0 and 1, blood will be collected for analysis. Further cognitive, quality of life and pain questionnaires will be administered perioperatively.

ELIGIBILITY:
Inclusion Criteria:

* Over 60 years of age
* Inpatient and scheduled for surgical procedure at MGH

Exclusion Criteria:

* Blindness, deafness or the inability to speak English
* Inability to provide informed consent

Objective Drop Criteria

* Post-operative intubation greater than 24 hours

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatients over the age of 60 scheduled for a surgical procedure at MGH
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ibala R, Mekonnen J, Gitlin J, Hahm EY, Ethridge BR, Colon KM, Marota S, Ortega C, Pedemonte JC, Cobanaj M, Chamadia S, Qu J, Gao L, Barbieri R, Akeju O. A polysomnography study examining the association between sleep and postoperative delirium in older hospitalized cardiac surgical patients. J Sleep Res. 2021 Oct;30(5):e13322. doi: 10.1111/jsr.13322. Epub 2021 Mar 24. PMID 33759264

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MGH Surgery Patients
Started | 38
Completed Baseline Assessment | 32
Completed PSG | 25
Completed | 17
Not Completed | 21
Not completed — Found Ineligible | 2
Not completed — Withdrawal by Subject | 14
Not completed — Lost to Follow-up | 4
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: 38 Patients enrolled in the study. 32 Patients completed the baseline assessment.
Arm/Group | MGH Surgery Patients
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants] — Based on number of patients who enrolled.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 4
    >=65 years | 34
Age, Continuous [Mean (Standard Deviation); unit: years] — Based on number of patients who enrolled.
  years | 72 (5.98)
Sex: Female, Male [Count of Participants; unit: Participants] — Based on number of patients who enrolled.
  Participants
    Female | 8
    Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Based on number of patients who completed the baseline assessment. Population: Based on number of participants who completed the baseline assessment. Ethnicity data was collected during the baseline assessment.
  Participants
    number analyzed (Participants) | 32
    Hispanic or Latino | 0
    Not Hispanic or Latino | 32
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Based on number of patients who completed the baseline assessment. Population: Based on number of participants who completed the baseline assessment. Race data was collected during the baseline assessment.
  Participants
    number analyzed (Participants) | 32
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 30
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Association Between Sleep and POD
Description: Duration of sleep in delirious vs non-delirious patients
Time Frame: Night before surgery, approximately 13 hours
Population: Many of the PSG data samples that were collected the night of surgery were not interpretable and poor quality.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | MGH Surgery Patients
Number analyzed (Participants) | 16
Minutes
  Non Delirium: number analyzed (Participants) | 9
  Non Delirium | 278.5 [239.5 to 315.5]
  Delirium: number analyzed (Participants) | 7
  Delirium | 313.5 [271.3 to 352.5]

2. Secondary Outcome: Burst Suppression Ratio
Description: Burst suppression ratio during cardiopulmonary bypass. EEG recordings from the operating room were collected and analyzed for burst suppression.
Time Frame: Length of surgery (2-12 hours)
Population: Only 14 EEG recordings were analyzed. EEG recordings for other patients were not analyzed due to poor quality or lack of recording due to electronic or manual error during surgery.
Measure: Median (Inter-Quartile Range); unit: ratio
Groups:
- MGH Surgery Patients: PSG and EEG data will be collected, and delirium assessments conducted, on patients undergoing surgery at MGH.
  PSG data to be collected on the night before surgery to establish level of preexisting sleep disturbance. EEG data to be collected in the Operating room during surgery.
Arm/Group | MGH Surgery Patients
Number analyzed (Participants) | 14
ratio
  Patients screened positive for delirium: number analyzed (Participants) | 6
  Patients screened positive for delirium | 0.11 [0.02 to 0.43]
  Patients screened negative for delirium: number analyzed (Participants) | 8
  Patients screened negative for delirium | 0.00 [0.00 to 0.03]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected form the time the patient was enrolled to the completion of the follow-up assessment at 30 days.
Description: This study is an observational study, not an interventional study. Thus, all adverse events patients encounter during this time period would not be related to the research study.
  Adverse events and other events were determined by regular chart review.
Arm/Group | MGH Surgery Patients
All-Cause Mortality (participants affected / at risk) | 1/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

LIMITATIONS AND CAVEATS:
The quality of many of the PSG recordings was poor and not interpretable. After patients enrolled, many withdrew at the time the PSG was to be placed. So, sleep was recorded for fewer patients. Blood was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT03498560/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT03498560/ICF_001.pdf